CLINICAL TRIAL: NCT06326333
Title: The Effects of Combination of PSB and SAPB on Postoperative Analgesia in Coronary Artery Bypass Graft Surgery
Brief Title: Combination of Parasternal and Serratus Anterior Plane Block in Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Nilgün Zengin, Principal İnvestigator, Ankara City Hospital Bilkent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E.Kurul-E2-24-6176
Record Dates: First submitted 2024-03-17; First posted 2024-03-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Parasternal Block; Serratus Anterior Plane Block; Acute Pain; Postoperative Analgesia; Cardiac Surgery
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined parasternal block and serratus anterior plane block (Other): In the parasternal block application, the needle will be advanced under the pectoralis major muscle and above the intercostal muscle with the ultrasound-guided in-plane technique. 7.5 ml of 0.25% bupivacaine will be injected into this area per each level, at the level of the second and fourth intercostal space.
  Then, in the serratus anterior plane block application, in the anterior axillary line, the needle will be advanced under the serratus anterior muscle, above the sixth rib, with the in-plane technique under ultrasound guidance. 10 ml of 0.25% bupivacaine will be injected into this area.
  The application will be applied bilaterally.
  Interventions: Procedure: Combined parasternal block and serratus anterior plane block

INTERVENTIONS:
Procedure: Combined parasternal block and serratus anterior plane block — The first PSB will be applied to the patients with 7.5 ml of 0.25% bupivacaine under real-time ultrasound guidance at the level of the second intercostal space.
  The second PSB will be applied to the patients with 7.5 ml of 0.25% bupivacaine under real-time ultrasound guidance at the level of the fourth intercostal space.
  The SAPB will be applied to the patients with 10 ml of 0.25% bupivacaine under real-time ultrasound guidance at the level of the sixth rib in the anterior axillary line.
  The block applications will be applied bilaterally.

SUMMARY:
Postoperative analgesia is a critical risk factor for the development of pulmonary and cardiovascular complications in coronary artery bypass graft (CABG) surgery. If patients with high pain levels cannot breathe effectively, it may lead to atelectasis, cardiac ischemia, and arrhythmias. This prolongs the time it takes for patients to be discharged and increases the frequency of postoperative pulmonary complications and postoperative morbidity.

In addition to intravenous medications, various neuraxial and peripheral nerve blocks can be used in cardiac surgery. In recent years, neuraxial anesthesia has been avoided due to the use of intraoperative high-dose heparin. As an alternative, peripheral nerve blocks have recently gained popularity. Parasternal block (PSB) and serratus anterior plane block (SAPB) are very superficial and easy to reach. Recently, in the literature, the number of cases performed with these blocks under ultrasound guidance and the number of randomized controlled prospective studies have increased.

With this study, it was aimed to observe the analgesic effects on both the sternum and the drain site by applying PSB and SAPB applications simultaneously in the postoperative analgesia of CABG patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old
* American Society of Anesthesiologists (ASA) physical status I-II-III
* BMI 18 to 30 kg/m2
* Elective coronary artery bypass graft (CABG) surgery

Exclusion Criteria:

* Patient refusing the procedure
* Emergency surgery
* History of chronic opioid or analgesic used

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Pain Scores | 0th hour of the extubation
  After the extubation, pain will be assessed for the sternum and the drain area at the 0th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 2nd hour of the extubation
  After the extubation, pain will be assessed for the sternum and the drain area at the 2nd-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 4th hour of the extubation
  After the extubation, pain will be assessed for the sternum and the drain area at the 4th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 8th hour of the extubation
  After the extubation, pain will be assessed for the sternum and the drain area at the 8th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 12th hour of the extubation
  After the extubation, pain will be assessed for the sternum and the drain area at the 12th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Remifentanyl Consumption | intraoperative period
  Remifentanyl consumption for intraoperative period will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Çankaya, Ankara, Turkey (Türkiye)